CLINICAL TRIAL: NCT03780712
Title: Neonatal Immune Dysfunction Associated to the Risk of Newborn Sepsis in Benin
Brief Title: Immune Dysfunction in Newborn Sepsis
Acronym: RECIPAL
Status: Completed | Type: Observational
Sponsor: BioMérieux (Industry)
Collaborators: Institut de Recherche pour le Developpement (Other Government); Centre National de la Recherche Scientifique, France (Other); IRCB (Institut de la Recherche Clinique du Bénin) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECIPAL
Record Dates: First submitted 2018-03-13; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Sepsis Newborn; Malaria; Immune Responses
MeSH Terms: conditions — Neonatal Sepsis; Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood heparin tube Whole blood PAXgene Whole blood EDTA Dry Blood Spot Faeces Ficoll processed mononuclear cells Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis Risk Group: 419 infants born from mothers at risk to deliver babies with neonatal infections in Cotonou hospitals (Benin) 166 infants without sepsis born from mothers enrolled in a study to monitor pregnancy-associated malaria and Intrauterine growth restriction in Benin
  Interventions: Other: Non applicable

INTERVENTIONS:
Other: Non applicable — No intervention as it is an observational study

SUMMARY:
The aim of the project is to study neonatal immune dysfunction associated to the risk of newborn sepsis in a malaria endemic area in Benin.

DETAILED DESCRIPTION:
The fetal immunological responses maturate gradually during the last 3 months of pregnancy. To respond to pathogens, newborns depend essentially on their innate immune system. Premature babies have a significant impairment of innate and immune regulatory functions, thus promoting neonatal sepsis. In addition, chronic infections during pregnancy, including those of parasitic origin, fetal immunity. In utero exposure to P. falciparum antigens impacts particularly the newborn immune development and is a risk factor predisposing to malaria and also to other infections during the first year of life.

The major objectives are to assess:

* The relevance of a host biomarker driven diagnostic of sepsis in newborns,
* The relevance of immune markers as indicators of sepsis incidence, secondary infections occurrence, and mortality
* The role of novel diagnostic techniques (FilmArray panels) as part of the microbiological diagnostic,
* The immunological profile of the infants in the 3 first months of life.

The targeted population is newborns with a high risk to develop sepsis recruited at delivery compared to a control infant population with a low infection risk.

ELIGIBILITY:
Inclusion Criteria for the sepsis risk group (400 infants):

* Child born from mothers having one of the following criteria before delivery will be included in this study:

  * Spontaneous preterm delivery (<37 weeks of gestation time)
  * Foul smelling / with meconium / colored / bloody amniotic liquid
  * Rupture of membranes > 18 hours
  * Maternal fever at delivery
  * Vaginal infection
* Child born at the maternity of CNHU (Centre National Hospitalier et Universitaire, Cotonou, Benin) or CHUMEL (Centre Hospitalier et Universitaire de la Mère et de l'Enfant Lagune, Cotonou, Benin) or HZAC (Hopital de zone d' Abomey-Calavi, Benin).
* Mother located near Abomey-Calavi. This criterion has been included to limit the follow-up expenses and spare the travel to the project staff in charge of the 3 month follow-up.

Inclusion Criteria for the control group (170 infants):

- Child born from mothers enrolled in the RECIPAL study (Pregnancy-associated malaria and Intrauterine growth restriction in Benin)

Exclusion Criteria for both groups:

* HIV + status or unknown HIV status of the mother (as the mother and child will be part of the national program to take care of mother and child HIV+ at delivery)
* Parents do not consent to be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The targeted population is newborns with a high risk to develop sepsis recruited at delivery compared to a control infant population with a low infection risk.
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2016-04-17 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Evaluate Procalcitonin (PCT) for early onset neonatal sepsis diagnostic | At birth
  To measure in cord blood the association and performance of PCT and the early diagnosis of neonatal sepsis for infants at risk to develop infection

SECONDARY OUTCOMES:
Evaluate Procalcitonin (PCT) for late onset neonatal sepsis diagnostic | At one week after birth
  To measure in peripheral blood the association and performance of PCT and the diagnosis of late onset neonatal sepsis for infants at risk to develop infection
To draw Procalcitonin (PCT) expression profile during 12 weeks after birth | Twelve weeks follow-up after birth
  To measure PCT concentration during 12 weeks (sampling at birth, week 1, week 4, week 8 and week 12) and explore the relevance of host biomarker-driven antibiotherapy in a low-income country
Evaluate 2 host biomarkers mRNA expression (CD74 and CX3CR1) to prognostic neonatal sepsis | Twelve weeks follow-up after birth
  To measure CD74 and CX3CR1 mRNA expression in order to evaluate their performance on the early prognostic of neonatal sepsis for infants at risk to develop infections (occurrence of secondary infections and mortality rate)
FilmArray panels for early diagnosis of neonatal sepsis | Twelve weeks follow-up after birth
  To test commercial FilmArray panels in order to evaluate the role of novel diagnostic techniques as part of the diagnostic algorithm on the early diagnosis of neonatal sepsis over a period of 12 weeks for infants at risk to develop infection

REFERENCES:
- [Derived] Ezinmegnon S, Mommert M, Bartolo F, Agbota G, Darius S, Briand V, d'Almeida M, Alao MJ, Dossou-Dagba I, Massougbodji A, Lausten-Thomsen U, Pachot A, Vachot L, Yugueros-Marcos J, Brengel-Pesce K, Fievet N, Tissieres P. Prospective multicentre study of host response signatures in neonatal sepsis in Sub Saharan Africa. Sci Rep. 2022 Dec 12;12(1):21458. doi: 10.1038/s41598-022-25892-x. PMID 36509812
- [Derived] Fievet N, Ezinmegnon S, Agbota G, Sossou D, Ladekpo R, Gbedande K, Briand V, Cottrell G, Vachot L, Yugueros Marcos J, Pachot A, Textoris J, Blein S, Lausten-Thomsen U, Massougbodji A, Bagnan L, Tchiakpe N, d'Almeida M, Alao J, Dossou-Dagba I, Tissieres P; SEPSIS study group collaborators; SEPSIS study group. SEPSIS project: a protocol for studying biomarkers of neonatal sepsis and immune responses of infants in a malaria-endemic region. BMJ Open. 2020 Jul 23;10(7):e036905. doi: 10.1136/bmjopen-2020-036905. PMID 32709653